CLINICAL TRIAL: NCT03086681
Title: A Multicenter, Randomized Controlled Clinical Trial Comparing Endostar With Concurrent Chemoradiotherapy Versus Concurrent Chemoradiotherapy in the Treatment of Locally Advanced Cervical Carcinoma
Brief Title: Endostar Combined With Concurrent Chemoradiotherapy For Locally Advanced Cervical Carcinoma
Acronym: ECWHCCFLACC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yong Zhang,MD (Other)
Responsible Party: Sponsor-Investigator, Yong Zhang,MD, MD, First Affiliated Hospital of Guangxi Medical University
Organization: First Affiliated Hospital of Guangxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FirstGuangxiMU-2016-062
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cervical Carcinoma
Keywords: Cervical carcinoma; endostar; concurrent chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — endostar protein; Endostatins; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- concurrent chemoradiotherapy + endostar (Experimental): 4 cycles of Endostar and 5 cycles of DDP concurrent with radiotherapy
  Interventions: Drug: Endostar; Drug: DDP
- concurrent chemoradiotherapy (Active Comparator): 5 cycles of DDP concurrent with radiotherapy
  Interventions: Drug: DDP

INTERVENTIONS:
Drug: Endostar — Endostar: 7.5mg/m2 d1-10, repeat every 15 days, for 4 cycles
  Other Names: recombinant human endostatin
  Arms: concurrent chemoradiotherapy + endostar
Drug: DDP — DDP: 40mg /m2，per week, for 5 cycles
  Other Names: cisplatin

SUMMARY:
A total of 120 patients with pathologically confirmed Locally advanced cervical carcinoma were enrolled. Patients were randomly divided into two groups, with 60 patients in each group. One group was treated with Concurrent Chemoradiotherapy combined with Endostar and the other group was treated with Concurrent Chemoradiotherapy. The short term efficacy and the toxic of these treatments were evaluated. The 1-year, 3-year, 5-year overall survival and progression-free survival of patients were analyzed. The investigators data may provide an alternative option for the treatment of Locally advanced cervical carcinoma with high efficacy and low toxicity.

DETAILED DESCRIPTION:
This study was a multicenter, randomized controlled clinical trial. A set of unified standards were used, including the clinical research program, inclusion criteria, exclusion criteria, chemoradiotherapy regimen and evaluation criteria. Nine medical centers participated in this study and 120 patients with pathologically confirmed Locally advanced cervical carcinoma were enrolled. These patients were randomly divided into two groups: concurrent chemoradiotherapy combined with Endostar group ( IMRT 45-50Gy, DDP 40mg/m2, per week for 5cycles, Endostar: 7.5mg/m2 d1-10, repeat every 15 days, for 4 cycles) and concurrent chemoradiotherapy group ( IMRT 45-50Gy, DDP 40mg/m2, per week, for 5cycles). After treatment, follow-up was performed every 3 months. The treatment toxicity, local control rate, distant metastasis-free survival, overall survival, progression-free survival were observed and assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients of either gender and aged from 18 to 65 years old.
* patients with histologically confirmed cervical carcinoma.
* patients at stage Ib, IIa2, IIb-IVa by FIGO 2009 staging.
* KPS ≥ 70 (Appendix I)
* patients with available MRI or CT data of cervical and measurable tumor lesions.
* patients did not receive any treatment before enrollment.
* patients with expected survival longer than 6 months.
* biochemical indexes: WBC > 4,000/mm3, and blood platelet ≥ 100,000 mm3; PT≤UNL; levels of indicators for hepatic and renal function was 1.5 folds of the upper limit of normal value.
* the informed content was obtained from every patient.
* patients with effective follow-up.

Exclusion Criteria:

* those with malignant tumors other than cervical carcinoma.
* those received treatments before enrollmment.
* lactating women and Pregnant woman.
* those who were undergoing other drug trials.
* those with severe complications, including myocardial infarction, severe arrhythmia, severe cerebrovascular disease, ulcer disease, mental illness and uncontrollable diabetes.
* those who were treated with tumor targeting drugs.
* those who could not subject to MRI or CT examination.
* those who could not meet the requirements of the prescribed dose.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
short-time effect | 3 months
  3 months after treatment, the subjects go into observation period. MRI/CT will be used for evaluating the carcinoma status.

SECONDARY OUTCOMES:
Overall Survival | 3 years,5 years
  OS was calculated from the date of entry into the study to the date of death or the last follow-up visit.
Progression-Free Survival | 3 years,5 years
  PFS was calculated from the date of entry into the study to the date of first physical or radio-graphic evidence of disease progression, death or the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Zhang, MD, Study Chair — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu F, Tang X, Liu W, Luo Z, Huang H, Liu M, Wang H, Liao S, Ma S, Jiang L, Zhang Y. Efficacy of Endostar plus concurrent chemoradiotherapy in locally advanced cervical cancer: a multicenter, phase II randomized trial. Ther Adv Med Oncol. 2025 Oct 3;17:17588359251379397. doi: 10.1177/17588359251379397. eCollection 2025. PMID 41049580
- See also: Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. — https://www.ncbi.nlm.nih.gov/pubmed/25651787
- See also: Improved survival with bevacizumab in advanced cervical cancer. N Engl J Med. 2014 Feb 20;370(8):734-43. doi: 10.1056/NEJMoa — https://www.ncbi.nlm.nih.gov/pubmed/24552320
- See also: Concurrent chemotherapy and pelvic radiation therapy compared with pelvic radiation therapy alone as adjuvant therapy after radical surgery in high-risk early-stage cancer of the cervix. J Clin Oncol 2000;18:1 — http://www.ncbi.nlm.nih.gov/pubmed/10764420
- See also: Pelvic radiation with concurrent chemotherapy compared with pelvic and para-aortic radiation for high-risk cervical cancer. N Engl J Med 1999;340:1137-1143. — http://www.ncbi.nlm.nih.gov/pubmed/10202164
- See also: Pelvic radiation with concurrent chemotherapy compared with pelvic and para-aortic radiation for high-risk cervical cancer. — http://www.ncbi.nlm.nih.gov/pubmed/10202164
- See also: Cisplatin, radiation, and adjuvant hysterectomy compared with radiation and adjuvant hysterectomy for bulky stage IB cervical carcinoma. — https://www.ncbi.nlm.nih.gov/pubmed/10202166
- See also: Concurrent cisplatin-based radiotherapy and chemotherapy for locally advanced cervical cancer — http://www.ncbi.nlm.nih.gov/pubmed/12109823
- See also: A randomized comparison of fluorouracil plus cisplatin versus hydroxyurea as an adjunct to radiation therapy in stages IIB-IVA carcinoma of the cervix with negative para-aortic lymph nodes — https://www.ncbi.nlm.nih.gov/pubmed/10334517
- See also: Survival and recurrence after concomitant chemotherapy and radiotherapy for cancer of the uterine cervix: a systematic review and meta-analysis — https://www.ncbi.nlm.nih.gov/pubmed/11564482
- See also: Clinical efficacy of modified preoperative neoadjuvant chemotherapy in the treatment of locally advanced (stage IB2 to IIB) cervical cancer: randomized study — https://www.ncbi.nlm.nih.gov/pubmed/18606439
- See also: Reducing uncertainties about the effects of chemoradiotherapy for cervical cancer: a systematic review and meta-analysis of individual patient data from 18 randomized trials — https://www.ncbi.nlm.nih.gov/pubmed/19001332
- See also: Modern radiotherapy and cervical cancer. — https://www.ncbi.nlm.nih.gov/pubmed/21053528
- See also: Quality of life (QOL) outcomes from a randomized trial of cisplatin versus cisplatin plus paclitaxel in advanced cervical cancer: a Gynecologic Oncology Group study — https://www.ncbi.nlm.nih.gov/pubmed/16376417
- See also: A randomized trial comparing concurrent chemoradiotherapy with single-agent cisplatin versus cisplatin plus gemcitabine in patients with advanced cervical cancer — https://www.ncbi.nlm.nih.gov/pubmed/25827291
- See also: Role of angiogenesis in tumor growth and metastasis — https://www.ncbi.nlm.nih.gov/pubmed/12516034
- See also: Antiangiogenic agents and their promising potential in combined therapy — http://www.ncbi.nlm.nih.gov/pubmed/11418313
- See also: Function of endogenous inhibitors of angiogenesis as endothelium specific tumor suppressors — http://www.ncbi.nlm.nih.gov/pubmed/15710885
- See also: Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung caner — http://www.ncbi.nlm.nih.gov/pubmed/17167137
- See also: Phase II trial of bevacizumab in the treatment of persistent or recurrent squamous cell carcinoma of the cerix: a gynecologic oncology group study — http://www.ncbi.nlm.nih.gov/pubmed/19139430
- See also: Incorporation of bevacizumab in the treatment of recurrent and metastatic cervical cancer: a phase III randomized trial of the Gynecologic Oncology Group — http://www.ncbi.nlm.nih.gov/pubmed/25842084
- See also: Clinical potential of bevacizumab in the treatment of metastatic and locally advanced cervical cancer — http://www.ncbi.nlm.nih.gov/pubmed/26418895